CLINICAL TRIAL: NCT01117753
Title: Stage II Research on Outpatient Treatment for Adolescents With Comorbidity
Brief Title: Research on Outpatient Adolescent Treatment for Comorbid Substance Use and Internalizing Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUSC19301; 1R01DA025616-01A1 (NIH)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2013-05

CONDITIONS: Substance-Related Disorders; Depressive Disorder; Anxiety Disorder
MeSH Terms: conditions — Substance-Related Disorders; Depressive Disorder; Anxiety Disorders | interventions — Ambulatory Care; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OPT-A (Experimental): OPT-A is an outpatient family-based treatment for co-occurring substance use and internalizing disorders
  Interventions: Behavioral: OutPatient Treatment for Adolescents (OPT-A)
- Treatment as Usual (Active Comparator): Treatment as usual in a community based mental health center
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: OutPatient Treatment for Adolescents (OPT-A)
  Arms: OPT-A
Behavioral: Treatment As Usual
  Arms: Treatment as Usual

SUMMARY:
Adolescent substance abuse results in significant negative outcomes and extraordinary costs for youths, their families, communities, and society. Moreover, rates of psychiatric comorbidity among substance abusing youth range from 25% up to 82%, and youths with a dual diagnosis are more than twice as costly to treat compared to those with no comorbidity. The applicant principal investigator recently completed a pilot project funded by the National Institute on Drug Abuse focused on developing and piloting a psychosocial treatment specifically for youth presenting for outpatient treatment with co-occurring substance use and internalizing (i.e., mood and/or anxiety) problems. Results were promising with the experimental group exhibiting significantly less substance use and more rapid reductions in anxiety and depressive symptoms compared to the control group. The proposed research is a randomized clinical trial (RCT) to compare the experimental treatment (OutPatient Treatment for Adolescents; OPT-A) to an "active placebo" on key clinical indices from pre-treatment through 18 months. The proposed RCT (n = 160) employs the treatment manual, quality assurance protocol, and therapist training protocol developed and successfully tested in the pilot study, to evaluate the efficacy of OPT-A for youth referred to outpatient treatment of co-occurring substance use and internalizing problems. The following outcomes will be evaluated: drug use; mental health; behavioral, school, peer, and family functioning; and consumer satisfaction. The intervention addresses one of the more prevalent and most challenging, costly, and understudied presenting problems among adolescent outpatients. If successful, this research could provide a considerable contribution in the treatment field for youth with co-occurring substance use and internalizing disorders.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 17 years of age
* Residing with at least one adult caregiver who serves as a parent figure
* In need of treatment for a Substance Abuse or Dependence Disorder
* In need of treatment for an Axis I Mood Disorder and/or Anxiety Disorder

Exclusion Criteria:

* Pervasive Developmental Disorder
* Active Psychotic Disorder
* Severe or profound mental retardation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Substance use | baseline and 1-, 2-, 3-, 6-, 12-, and 18-month follow-up
Mental Health | baseline and 1-, 2-, 3-, 6-, 12-, and 18-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ashli J Sheidow, PhD, Principal Investigator — Medical University of South Carolina, Department of Psychiatry & Behavioral Sciences, Family Services Research Center
Locations (1):
- Medical University of South Carolina, Department of Psychiatry & Behavioral Sciences, Family Services Research Center, Charleston, South Carolina, United States